CLINICAL TRIAL: NCT01007630
Title: A Prospective Randomized Placebo-Controlled Double-Blind Study Assessing Change in Olfactory Function After Initiation of Rasagiline in Idiopathic Parkinson's Disease
Brief Title: A Study Assessing Change in Sense of Smell After Rasagiline Use in Parkinson's Patients
Acronym: PD-SOAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Parkinson's Institute (Other)
Collaborators: Teva Neuroscience, Inc. (Industry)
Responsible Party: Principal Investigator, Grace Liang, Principal Investigator, Director of Clinical Trials, The Parkinson's Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD-SOAR
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; Parkinsons; Parkinson; Parkinson's Disease; PD; Rasagiline; Azilect; Olfactory; Sense of Smell; UPSIT
MeSH Terms: conditions — Parkinson Disease; Anosmia | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline (Active Comparator): 0.5mg of Rasagiline for 14 days, then switch to 1mg of Rasagiline for remainder of the study (approximately 10 weeks total).
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): 0.5mg of placebo for 14 days, then switch to 1mg of placebo for remainder of the study (approximately 10 weeks total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — 0.5mg for 14 days, then switch to 1mg for remainder of the study (approximately 10 weeks total)
  Other Names: Brand Name: Azilect
  Arms: Rasagiline
Drug: Placebo — 0.5mg for 14 days, then switch to 1mg for remainder of the study (approximately 10 weeks total)
  Arms: Placebo

SUMMARY:
A decrease or loss of the sense of smell is very common in patients with Parkinson's Disease even in the earliest stages of the disease. There have been no treatments that have been proven to improve sense of smell in patients with Parkinson's Disease.

Rasagiline (brand name: Azilect) was approved by the U.S. Food and Drug Administration (FDA) on May 16th 2006 to be used by Parkinson's patients to treat the motor symptoms associated with the disease. The purpose of this study is to see if there is change in sense of smell after starting Rasagiline.

DETAILED DESCRIPTION:
This study will last approximately 10 weeks.

* 2 visits to The Parkinson's Institute in Sunnyvale, California
* 1 phone call between visits

You will be asked to take either Rasagiline (Azilect) or placebo (an identical pill without active ingredients)

* 5 in 6 chance of receiving Rasagiline (Azilect)
* 1 in 6 chance of receiving placebo
* Neither you nor the study team will know which you are assigned
* This information will be available in case of emergency

To be eligible for this study, you must:

* be 90 years old or younger
* have a decreased loss of smell or complete loss of smell
* have not taken Selegiline or Rasagiline within the past 12 months
* have not smoked within the last year
* be on a stable dose of Parkinson's medication (or not on any PD medicines)
* have no history of head trauma, nasal surgery, nasal inflammation causing congestion or polyps, nasal/sinus infection, or prior Zicam use
* have not used decongestants, antihistamine or inhaled steroids within 2 weeks of the study and be willing to avoid such treatments during the study

ELIGIBILITY:
Inclusion Criteria:

* Men and women with Parkinson's Disease (PD), defined as the presence of at least two of the cardinal signs of PD (bradykinesia, resting tremor, rigidity) without other identifiable cause of parkinsonism or signs of atypical parkinsonism
* Functional hyposmia or anosmia, as defined by UPSIT scores less than the 25th percentile for age- and gender-matched norms
* Have been on stable dose of PD medications for at least 30 days
* Age < or = 90 years
* Willing and able to give informed consent
* Women of child-bearing potential may participate provided they are willing to use adequate contraceptive methods during the duration of the study. Women of childbearing potential must have a negative pregnancy test at the screening visit and be non-lactating.

Exclusion Criteria:

* Prior use of an MAO inhibitor, including selegiline or rasagiline within the last 12 months
* Presence of other conditions that in the investigator's opinion may significantly cause olfactory impairment, including prior head trauma, nasal surgery, nasal inflammation causing concurrent congestion or polyps, nasal or sinus infection, prior intranasal zinc salt (Zicam) use, history of smoking within the past year
* Presence of dementia or significant cognitive impairment with Mini-Mental State Examination (MMSE) < 24
* Present of a medical or surgical condition which in the opinion of the investigator would preclude participation in and completion of study procedures
* Use of any experimental medication within 60 days of baseline
* Use of decongestants, antihistamines, inhaled steroids within 2 weeks of baseline
* Use of any medication contraindicated with use of rasagiline (Investigator will take into consideration concomitant antidepressant use as per prescribing information guidelines for rasagiline)

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in UPSIT score at 10-week visit | 10 weeks

SECONDARY OUTCOMES:
Tolerability: Number of subjects (%) who discontinue the study due to AEs | 10 weeks
Safety: AE incidence | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Liang, MD, Principal Investigator — The Parkinson's Institute
Locations (1):
- The Parkinson's Institute, Sunnyvale, California, United States

REFERENCES:
- See also: The Parkinson's Institute Clinical Trials Website — http://thepi.org/index.php?submenu=clinical_trials&src=gendocs&ref=ClinicalTrialsMain&category=clinical_trials